CLINICAL TRIAL: NCT06298669
Title: Selection of Cardiac Resynchronization Therapy Pacing Modalities in Patients Supported by LVADs
Brief Title: Biventricular Versus Right Ventricular Pacing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Coordinator support was lost
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Maya Guglin, Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 16052
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
Keywords: Left Ventricular Assist Device (LVAD); Cardiac resynchronization therapy (CRT)
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Biventricular Pacing followed by Right Ventricular Pacing (Experimental): Subjects will be randomly assigned to the order of pacing interventions. After baseline testing (with their CRT device still in the subjects' baseline pacing modality), subjects assigned to BiV-first will have their CRT device reprogrammed to BiV pacing modality in the clinic. After undergoing three months of treatment in this pacing modality, they will return to clinic for retesting. The CRT device will then be reprogrammed to RV pacing for the next 3 months. Subjects will then again return to clinic for retesting, and their CRT device will be reprogrammed to their baseline pacing modality.
  Interventions: Device: Biventricular Pacing; Device: Right Ventricular Pacing
- Right Ventricular Pacing followed by Biventricular Pacing (Experimental): Subjects will be randomly assigned to the order of pacing interventions. After baseline testing (with their CRT device still in the subjects' baseline pacing modality), subjects assigned to RV-first will have their CRT device reprogrammed to RV pacing modality in the clinic. After undergoing three months of treatment in this pacing modality, they will return to clinic for retesting. The CRT device will then be reprogrammed to BiV pacing for the next 3 months. Subjects will then again return to clinic for retesting, and their CRT device will be reprogrammed to their baseline pacing modality.
  Interventions: Device: Biventricular Pacing

INTERVENTIONS:
Device: Biventricular Pacing — The CRT device will be reprogrammed to coordinate contractions of the left and right ventricles.
Device: Right Ventricular Pacing — The CRT device will be reprogrammed for right ventricular contractions.
  Arms: Biventricular Pacing followed by Right Ventricular Pacing

SUMMARY:
The study is a randomized, single-blind crossover prospective study in which investigators will determine the clinical outcomes of cardiac resynchronization therapy (CRT) pacing modalities in patients with left ventricular assist devices (LVAD). Only patients are blinded. This is a small-scale study from which future larger scale randomized controls can be performed. The primary endpoint will be the effect of BiV and RV pacing setting on the 6-minute walk test.

DETAILED DESCRIPTION:
Heart failure patients with reduced left ventricular systolic function and worsening clinical status are frequently treated with mechanical devices. Cardiac resynchronization therapy (CRT) and left ventricular assist devices (LVAD) are mainstays of advanced heart failure treatment and have independently been demonstrated to decrease mortality. However, minimal research documents the utility of these two modalities in unison. There have been recent investigations comparing Biventricular (BiV) versus right ventricular (RV) pacing suggesting better exercise performance and decreased left ventricular (LV) volumes with RV pacing. This discovery contrasts with prior meta-analysis that reports no difference between LVAD patients with and without CRT including mortality and hospitalizations. Investigators aim to compare BiV pacing and RV pacing in LVAD patients with CRT on patient's exercise tolerance and frequency of tachyarrhythmias. Additionally, research is required to form a conclusion on the role of CRT in LVAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with both an LVAD and CRT device with functional leads
* Age 18 years and older
* Ability to walk
* Ability to sign consent

Exclusion Criteria:

* Patients with permanent atrial fibrillation
* Patients who are pacemaker dependent
* Patients with sustained ventricular tachycardia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (Three Months)
Arm/Group | Biventricular Pacing Followed by Right Ventricular Pacing | Right Ventricular Pacing Followed by Biventricular Pacing
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Period: Second Intervention (Three Months)
Arm/Group | Biventricular Pacing Followed by Right Ventricular Pacing | Right Ventricular Pacing Followed by Biventricular Pacing
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated after only one participant was enrolled in the study.
Arm/Group | Biventricular Pacing Followed by Right Ventricular Pacing
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Age is not reported for the single study participant to protect confidentiality.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Test Performance
Description: The distance walked over 6 minutes was measured at the baseline visit and the visit three months after baseline. The six month visit did not occur because the study was terminated.
Time Frame: Baseline visit; Three-month visit
Measure: Number; unit: meters
Arm/Group | Biventricular Pacing Followed by Right Ventricular Pacing
Number analyzed (Participants) | 1
meters
  Baseline visit | 350
  Three month visit | 375

2. Secondary Outcome: EQ-5D-3L Quality of Life Score
Description: Quality of Life was measured using the EQ-5D-3L questionnaire. The EQ-5D-3L asks participants to rate the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is rated as either no problems (score of 1), some problems (score of 2), or extreme problems (score of 3). Higher scores indicating a poorer overall quality of life in these dimensions. Scores on the five dimensions are summarized to create an index score. The EQ-5D-3L index score is a numerical value that summarizes a person's health state on a scale from -0.594 to 1:
  * 1: Full health
  * 0 or less: Equivalent to being dead or worse than dead
  The questionnaire was only completed at the baseline visit for the single participant on study.
Time Frame: Baseline visit
Measure: Number; unit: score on a scale
Arm/Group | Biventricular Pacing Followed by Right Ventricular Pacing
Number analyzed (Participants) | 1
score on a scale | -0.293

3. Secondary Outcome: Serum NT-PRO-BNP
Description: Serum levels of N-terminal pro-brain natriuretic peptide (NT-PRO-BNP) were measured at the baseline visit and the visit three months after baseline. The six month visit did not occur because the study was terminated.
Time Frame: Baseline visit; Three-month visit
Measure: Number; unit: pg/mL
Arm/Group | Biventricular Pacing Followed by Right Ventricular Pacing
Number analyzed (Participants) | 1
pg/mL
  Baseline visit | 470
  Three-month visit | 515

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Biventricular Pacing Followed by Right Ventricular Pacing
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT06298669/Prot_SAP_000.pdf